CLINICAL TRIAL: NCT05372718
Title: Multicenter, Open-label, Randomized Clinical Trial of Efficacy and Safety of the Thrombolysis With Recombinant Non-immunogenic Staphylokinase (Fortelyzin®) in Patients With ALI vs Surgery
Brief Title: Thrombolysis With Recombinant Non-immunogenic Staphylokinase vs Surgery in Patients With Acute Limb Ischemia FORAT Trial
Acronym: FORAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Supergene, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORAT
Record Dates: First submitted 2022-04-28; First posted 2022-05-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Acute Limb Ischemia
Keywords: acute limb ischemia; thrombolysis; thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Intervention Model Description: At clinical centers, patients will be randomly distributed by the "envelope method" into two groups for assignation Fortelyzin® or surgical methods of treatment.
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant non-immunogenic staphylokinase (Experimental): lyophilisate for preparation a solution, 5 mg (745,000 IU) in 20 ml over 1 minute through a perforated multihole catheter intrathrombally.
  30 minutes after this injection, infusion of recombinant non-immunogenic staphylokinase will be continued at a dose of 1 mg/hour, maximum 10 mg (50 ml) for 10 hours through a perforated multihole catheter intrathrombally.
  Interventions: Drug: Recombinant non-immunogenic staphylokinase (Fortelyzin®)
- Surgical methods of treatment (Experimental): endovascular intervention, open surgery and/or bypass surgery in accordance with the current National Guidelines
  Interventions: Procedure: surgical methods of treatment

INTERVENTIONS:
Drug: Recombinant non-immunogenic staphylokinase (Fortelyzin®) — lyophilisate for preparation a solution
  Other Names: Fortelyzin®
  Arms: Recombinant non-immunogenic staphylokinase
Procedure: surgical methods of treatment — Endovascular intervention, open surgery and/or bypass surgery in accordance with the current National Guidelines
  Arms: Surgical methods of treatment

SUMMARY:
Objective: to evaluate the efficacy and safety of intra-arterial intrathrombus administration of the recombinant non-immunogenic staphylokinase (Fortelyzin®) in patients with acute limb ischemia (ALI) vs surgery.

DETAILED DESCRIPTION:
Fortelyzin® (the active substance Forteplase) is a recombinant non-immunogenic staphylokinase with high fibrinselective thrombolytic activity. In a multicentre, randomised clinical trial in patients with ST-segment elevation myocardial infarction (FRIDOM), non-immunogenic staphylokinase was administered as a single intravenous bolus of 15 mg in all patients, regardless of bodyweight, and showed similar high reperfusion patency and fewer minor bleeding events compared with tenecteplase, as well as the absence of neutralising IgGs. Results of the multicentre, randomised clinical trial in patients with an acute ischaemic stroke (FRIDA) suggested that the non-immunogenic staphylokinase administrated as a single intravenous bolus of 10 mg in all patients within the 4-5 h after the onset of symptoms is non-inferior to alteplase. Mortality, symptomatic intracranial haemorrhage, and serious adverse events did not differ between treatment groups.

Mortality in the ALI continues to be high. According to the Guidelines on the management of patients with ALI, intravenous systemic thrombolysis is ineffective in patients with this condition. In contrast, catheter-directed thrombolysis based on the principle that activation of fibrin-bound plasminogen to the active enzyme plasmin is the most effective approach of lysing pathologic thrombi in the lower extremities of I-II b degree of ALI (Evidence level I-A).

So the main objective of this study is to evaluate the efficacy and safety of intra-arterial intrathrombus administration of the recombinant non-immunogenic staphylokinase (Fortelyzin®) in patients with ALI vs surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and older;
* Diagnosis of I-II b degree of ALI;
* Patient consent to use reliable contraceptive methods throughout the study and for 3 weeks after:

  * women who have a negative pregnancy test and use the following contraceptives: intrauterine devices, oral contraceptives, contraceptive patch, prolonged injectable contraceptives, double barrier method of contraception. Women who are not fertile can also take part in the study (documented conditions: hysterectomy, tubal ligation, infertility, menopause for more than 1 year);
  * men using barrier contraception. The study may also involve men who are not fertile (documented conditions: vasectomy, infertility);
* Availability of signed and dated informed consent of the patient to participate in the study.

Exclusion Criteria:

* Extensive bleeding at present;
* Intracranial (including subarachnoid) hemorrhage at present;
* Recent gastrointestinal bleeding (within 10 days);
* Major surgery or major trauma within the previous 3 months, recent traumatic brain injury;
* Systolic blood pressure above 180 mm Hg or diastolic blood pressure above 110 mm Hg or the need for intravenous drugs to lower blood pressure to these limits;
* Pregnancy, lactation;
* Known hypersensitivity to Fortelyzin®;
* Platelet count less than 100,000/µL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients without amputations | 30 days post randomization
  Outcome Measure is evaluated in terms of the number of patients without amputations

OTHER OUTCOMES:
Safety endpoint - Death from all causes | 30 days post randomization
  The safety is evaluated in terms of the number of deaths from all causes
Safety endpoint - hemorrhagic stroke | 30 days post randomization
  The safety is evaluated in terms of the number of hemorrhagic stroke
Safety endpoint - BARC type 3 and 5 bleeding | 30 days post randomization
  The safety is evaluated in terms of the number of BARC type 3 and 5 bleeding
Safety endpoint - Number and severity of serious adverse events (SAEs) and AEs in organs and systems | 30 days post randomization
  The safety is evaluated in terms of the number and severity of SAEs and AEs in organs and systems

CONTACTS AND LOCATIONS:
Overall Officials: Igor I. Zatevakhin, MD, PhD, Principal Investigator — N.I. Pirogov Russian Medical University, President of the Russian Society of Surgeons; Sergey S. Markin, MD, PhD, Study Director — Supergene, LLC
Locations (8):
- Russia (8):
  - Kursk city emergency hospital, Kursk, Kursl Region
  - Sergiyev Posad Regional Clinical Hospital, Sergiyev Posad, Moscow Oblast
  - Kaliningrad Regional Clinical Hospital, Kaliningrad
  - Kazan City Hospital No. 7, Kazan'
  - S.S. Yudin City clinical hospital, Moscow
  - S.P. Botkin Moscow Multidisciplinary Scientific and Clinical Center, Moscow
  - Ufa Emergency City Hospital, Ufa
  - Volgograd City Clinical Hospital of Emergency #25, Volgograd

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gusev EI, Martynov MY, Nikonov AA, Shamalov NA, Semenov MP, Gerasimets EA, Yarovaya EB, Semenov AM, Archakov AI, Markin SS; FRIDA Study Group. Non-immunogenic recombinant staphylokinase versus alteplase for patients with acute ischaemic stroke 4.5 h after symptom onset in Russia (FRIDA): a randomised, open label, multicentre, parallel-group, non-inferiority trial. Lancet Neurol. 2021 Sep;20(9):721-728. doi: 10.1016/S1474-4422(21)00210-6. PMID 34418399